CLINICAL TRIAL: NCT07218978
Title: Ripe for Revival: Outcomes Evaluation of a Mobile Produce Market With Vouchers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina State University (Other)
Collaborators: East Carolina University (Other)
Responsible Party: Principal Investigator, Basheerah Enahora, Assistant Professor, North Carolina State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 28013
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Diet Interventions; Food Security; Nutrition Security; Fruit and Vegetable Intake
Keywords: Mobile market; Lower-income; Fruit and Vegetable Intake; Quasi-Experimental; Vouchers; Nutrition Incentives

STUDY DESIGN:
Intervention Model Description: Quasi-experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Voucher Recipients (Experimental): Voucher participants will be referred by Extension professionals who serve lower-resourced individuals during routine programs
  Interventions: Behavioral: Mobile Market Voucher Outcomes Study

INTERVENTIONS:
Behavioral: Mobile Market Voucher Outcomes Study — Voucher participants will be referred by Extension professionals who serve lower-resourced individuals during routine programs (i.e., NC Extension programs such as Expanded Food and Nutrition Education Program (EFNEP). After receiving the referrals from Extension professionals, a member of the research team will contact the referred participant to provide a $20 monthly voucher for three months for use at the mobile market. Trained researchers will collect data at baseline (when a voucher is issued), at ~4 weeks (2nd voucher), 8 weeks (3rd voucher) and 12-16 weeks (post-program) at the NC Cooperative Extension office. FV intake will be measured by skin carotenoid scan. Researchers will obtain height (baseline), weight, and blood pressure at each data collection time point. Survey measures will include the secondary outcomes using adapted versions of validated instruments, with questions on demographics, and food and nutrition security status.

SUMMARY:
Increasing access to healthy foods is crucial to combating chronic disease in rural communities. The Ripe for Revival mobile market, a non-profit eastern NC-based mobile market, seeks to improve healthy food access among those at greatest risk of food insecurity and poor health. By implementing vouchers at the mobile market, this study will help make healthy food affordable and accessible. This project is poised to improve diet and health among rural residents in eight counties and promote sustainable local food systems in North Carolina.

DETAILED DESCRIPTION:
Increasing fruit and vegetable (FV) intake and reducing saturated fat, salt, and added sugar are central lifestyle recommendations in the Dietary Guidelines for Americans to prevent chronic disease. Yet, while diet is modifiable, rural families face structural and systemic inequities that make accessing affordable, healthy food more difficult.

Recognizing these disparities and adverse impacts, there is a clear need to create opportunities for improved nutrition through comprehensive solutions that account for rurality, affordability, and accessibility. One potential strategy to improve rural food access is mobile markets. Ripe for Revival is a 501(c)3 based in Rocky Mount, North Carolina, with a mission to increase access to fresh foods in lower-resourced communities with a mobile market model. Ripe for Revival owns and operates a produce farm, purchases excess food from eastern NC farmers, and then sells fresh foods to patrons at roughly 20% discounted prices through its mobile market. The mobile market (a retrofitted school bus) offers fresh produce, eggs, meat, and milk weekly in eastern and central NC counties This project continues NC State Extension's partnership with Ripe for Revival to implement vouchers to help increase mobile market affordability and assess program impacts among rural NC families. The specific aims of this proposed study include:

Aim 1. Determine the nutrition-related impacts of mobile market vouchers among Ripe for Revival patrons in six rural eastern NC counties (Bertie, Halifax, Hertford, Lenoir, Northampton, and Washington).

Aim 2. Examine voucher redemption rates, volume and dollars of local produce purchased, and suggestions for mobile market improvements among Ripe for Revival mobile market customers.

This proposed project will promote health and advance equity among underserved rural families. The project addresses barriers to equitable food access, promotes a balanced diet to prevent chronic disease, and fosters sustainable local agriculture through a mobile market model.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Communicates fluently in English or Spanish
* An active participant in an NC Cooperative Extension program May 2025 - June 2027
* At risk of food insecurity
* Willing to shop at or visit a Ripe for Revival mobile produce market
* Willing to use the provided $20 monthly voucher to shop at the Ripe for Revival mobile produce market
* Works or lives in a North Carolina county where this study is being conducted, including Bertie, Halifax, Hertford, Jones, Lenoir, Northampton, Warren, or Washington

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria above cannot participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Skin Carotenoids | Enrollment/baseline (week 0), 4 weeks, 8 weeks and at 12-16 weeks
  Fruit and vegetable intake measured by skin carotenoids (derived from a validated reflection spectroscopy device, Veggie Meter®

SECONDARY OUTCOMES:
Fruit and vegetable intake | Enrollment/baseline (week 0), 4 weeks, 8 weeks and at 12-16 weeks
  Measured by DSQ FV Module - GusNIP NTAE Survey
Weight/Body Mass Index | Enrollment/baseline (week 0), 4 weeks, 8 weeks and at 12-16 weeks
  Weight/Body Mass Index. Weight measured by electronic scale with standiometer SECA 874 as the average of two measures. Height (baseline only).
Blood Pressure | Enrollment/baseline (week 0), 4 weeks, 8 weeks and at 12-16 weeks
  Blood pressure measured by noninvasive automated monitor (Omron HEM-907XL, Vernon Hills, IL) with a first measure after seated for 5 minutes and 2 repeat measures at 1-minute intervals.
Food Security Status | Enrollment/baseline (week 0), 4 weeks, 8 weeks and at 12-16 weeks
  Food security status measured by USDA household 6-item screener
Nutrition Security Status | Enrollment/baseline (week 0), 4 weeks, 8 weeks and at 12-16 weeks
  Measured by the Center for Nutrition & Health Impact 4-item Nutrition Security Screener
Food Utilization | Enrollment/baseline (week 0), 4 weeks, 8 weeks and at 12-16 weeks
  Measured by the Center for Nutrition & Health Policy Impact 4-item screener
Voucher Redemption Rate | Enrollment/baseline (week 0), 4 weeks, 8 weeks and at 12-16 weeks
  Measured by Mobile Market POS system
Pounds of produce/local produce volume | Enrollment/baseline (week 0), 4 weeks, 8 weeks and at 12-16 weeks
  Measured by mobile market POS system
Mobile Produce Market Satisfaction | Enrollment/baseline (week 0), 4 weeks, 8 weeks and at 12-16 weeks
  Measured by self-reported survey

CONTACTS AND LOCATIONS:
Overall Officials: Basheerah Enahora, PhD, RDN, LDN, Principal Investigator — NC State University
Locations (1):
- NC State University, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Researchers will not make individual participant data available. Researchers will share aggregated participant results